CLINICAL TRIAL: NCT04945369
Title: Follow-up During the Peripubertal Period of Preterm Children (Under 35 Weeks of Amenorrhea) Included in the "EPIPOD" Protocol : Evaluation of Insulin Resistance
Brief Title: Follow-up During the Peripubertal Period of Preterm Children Included in the Protocol Entitled "EPIPOD".
Acronym: INFANTPOD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: RC20_0522
Record Dates: First submitted 2021-06-15; First posted 2021-06-30 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Preterm Children
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Children born prematurely included in the EPIPOD protocol and now in the peripubertal period (Experimental): At inclusion in the INFANTPOD study :
  * Blood and urinary samples collection for evaluation of insulin resistance and of renal function analysis.
  * Assessment of body composition by a commercialized device called "BOP-POD" and by impedancemetry
  * Assessment of pulse wave by a commercialized device called "popmetre"
  * Questionnaires for analysis of eating behaviour
  * Assessment of physical activity by a commercialized device called "accelerometer" and by questionnaire.
  Interventions: Other: clinical and biological measurements and questionnaires

INTERVENTIONS:
Other: clinical and biological measurements and questionnaires — Blood and urinary samples collection for evaluation of insulin resistance and of renal function analysis.
  Assessment of body composition by BOP-POD and by impedancemetry. Assessment of pulse wave by popmetre. Assessment of physical activity by accelerometer and by questionnaire Questionnaires for analysis of eating behaviour

SUMMARY:
Prematurity is associated with an increased risk of developing cardiovascular and metabolic disturbances in adulthood.

It has been demonstrated that the body composition of children born prematurely is different from that of children born under term with a deficit in fat free mass.

It can thus be wondered if this excessive adiposity does or does not predict the risk of insulin resistance in adulthood.

Children born prematurely, with a body composition measurement performed at discharge from neonatal hospitalization as part of the EPIPOD protocol, and now aged between 8 and 14 years, will be included in the INFANTPOD protocol.

Analysis of body composition, insulin resistance, renal function, pulse wave velocity, eating behaviour and of physical activity will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Children hospitalised at the Nantes University Hospital in the neonatal period
* With a body composition measurement performed at discharge from neonatal hospitalization as part of the EPIPOD protocol
* Born prematurely (under 35 weeks of amenorrhea)
* Included in the Lift cohort with follow-up up to 7 years
* Aged between 8 and 14 years at inclusion

Exclusion Criteria:

* Children with an isolated metabolic disease: insulin-dependent diabetes; endocrine disease (Cushing's, hypothyroidism)
* Age of 15 years or more
* with a chromosomal anomaly
* with contraindicating measurement of the BOP-POD: ventilatory support, continuous parenteral feeding, elimination stoma
* Refusal of either parent or child

Ages: 8 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 114 (Estimated)
Dates: Start 2022-02-02 (Actual); Primary Completion 2028-02-02 (Estimated); Study Completion 2028-02-02 (Estimated)

PRIMARY OUTCOMES:
Insulin resistance as measured by the Triglyceride-Glucose Index | 1 day

SECONDARY OUTCOMES:
Insulin resistance as measured by the Homeostasis Model Assessment - Insulin Resistance index | 1 day
Body composition (percentage of fat versus fat free mass) by BOP-POD and by impedancemetry (biodyXpert) for assessment of body composition variations between peripubertal period and neonatal period | 1 day
creatinine clearance | 1 day
Eating behaviour using standardized questionnaire named Child Eating Behaviour questionnaire | 1 day
Eating behaviour using standardized french questionnaire named "QCAJE Questionnaire Comportement Alimentaire du Jeune Enfant" | 1 day

CONTACTS AND LOCATIONS:
Locations (1):
- Nantes University Hospital, Nantes, France